CLINICAL TRIAL: NCT05605002
Title: Efficacy and Safety of Intradermal Acupuncture for Major Depressive Disorder: a Study Protocol for a Multicenter, Prospective, Randomized Controlled Trial
Brief Title: Efficacy and Safety of Intradermal Acupuncture for Major Depressive Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xiaomei Shao (Other)
Collaborators: Zhejiang Provincial Tongde Hospital (Other); First People's Hospital of Hangzhou (Other); The First Affiliated Hospital of Zhejiang Chinese Medical University (Other)
Responsible Party: Sponsor-Investigator, Xiaomei Shao, Professor, The Third Affiliated hospital of Zhejiang Chinese Medical University
Organization: The Third Affiliated hospital of Zhejiang Chinese Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022ZX010-INM
Record Dates: First submitted 2022-08-31; First posted 2022-11-03 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder; Intradermal Acupuncture; Magnetic Resonance Imaging
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Selective Serotonin Reuptake Inhibitors

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Waiting list group (Active Comparator): This group will include 30 patients with MDD who will be treated with oral SSRIs only, the dosage of which will be determined by the psychiatrist. After 6 weeks, patients could choose 6 weeks' intradermal acupuncture treatments free of charge.
  Interventions: Drug: SSRIs
- SIA+SSRIs group (Sham Comparator): This group will include 30 patients with MDD who will be treated with sham intradermal acupuncture combined with SSRIs. Acupoints related to MDD will be stimulated by acupuncturists and the dosage of oral SSRIs will be determined by the psychiatrist.
  Interventions: Drug: SSRIs; Procedure: SIA
- AIA+SSRIs group (Experimental): This group will include 30 patients with MDD who will be treated with active intradermal acupuncture combined with SSRIs. Acupoints related to MDD will be stimulated by acupuncturists and the dosage of oral SSRIs will be determined by the psychiatrist.
  Interventions: Drug: SSRIs; Procedure: AIA

INTERVENTIONS:
Drug: SSRIs — SSRIs antidepressants, including fluoxetine, paroxetine, sertraline, citalopram, etc., will be administered at oral doses determined by the psychiatrist. Once daily for 6 weeks.
  Other Names: selective 5-hydroxytryptamine reuptake inhibitors
Procedure: SIA — This study will select 4 acupoints (all taken bilaterally) commonly used to treat MDD, namely Taichong (LR3), Neiguan (PC6), Sanyinjiao (SP6) and Shenmen (HT7). The SIA will use the same size, colour and material as the AIA with a thin silicone pad in the middle instead of the needle body. SIA will be attached to the acupoints and retained for 72 hours, removed and rested for one day. A total of 10 sessions will be performed over a period of 6 weeks.
  Other Names: sham intradermal acupuncture
  Arms: SIA+SSRIs group
Procedure: AIA — This study will select 4 acupoints (all taken bilaterally) commonly used to treat MDD, namely Taichong (LR3), Neiguan (PC6), Sanyinjiao (SP6) and Shenmen (HT7). Depending on acupoints' location, a φ0.20*1.5mm or φ0.20*1.2mm AIA will be selected. Press the AIA to insert it vertically into the acupoint and retain it in the skin. AIA will be retained for 72 hours with a day's rest after removal. During the period of needle retention, participants will be instructed to press the AIA 3-4 times a day for approximately 1 minute each time, with as much stimulation as the patient can tolerate, at intervals of approximately 4 hours. A total of 10 sessions will be performed over a period of 6 weeks.
  Other Names: active intradermal acupuncture
  Arms: AIA+SSRIs group

SUMMARY:
Major depressive disorder (MDD) is a common mental illness that severely affects the health and quality of life of patients. Treatment with acupuncture alone or a combination of appropriate adjuncts has been reported to be significantly effective in reducing the severity of MDD, relieving patients' somatic symptoms and improving sleep. This study will focus on the intradermal acupuncture, which is more convenient, gentler and has longer lasting effects. The aim is to study the efficacy and safety of intradermal acupuncture for MDD, and to preliminarily explore the central nervous mechanisms by which it exerts its therapeutic effects.

DETAILED DESCRIPTION:
A total of 90 patients with MDD who meet the inclusion criteria will be included in the study. Participants will be randomly assigned 1:1:1 to the waiting list group (patients in this group will be treated with selective 5-hydroxytryptamine reuptake inhibitors (SSRIs) only), sham intradermal acupuncture combined with SSRIs (SIA) group and active intradermal acupuncture combined with SSRIs (AIA) group. The study will assess the efficacy and safety of intradermal acupuncture for MDD and examine whether intradermal acupuncture reduces side effects and improves the efficacy of SSRIs for MDD. In addition, the study will use magnetic resonance imaging (MRI) to study the possible central mechanisms by which intradermal acupuncture exerts its antidepressant effects.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with MDD according to the International Classification of Disease-10 (ICD-10);
2. Aged between 18 and 60 years (no limitation on gender);
3. No depression-related treatment in the past two weeks, except SSRIs;
4. Patients undergoing MRI and MRS should be right-handed and free of traumatic brain injury, claustrophobia or metal implants;
5. Written informed consent is obtained by the person or guardian.

Exclusion Criteria:

1. ICD-10 diagnoses: schizophrenia, bipolar disorder, manic episode or other psychotic disorders; alcohol and drug addiction;
2. Significant skin lesions, severe allergic diseases, tumors, and severe or unstable internal diseases involving the cardiovascular, digestive, endocrine, or hematological system;
3. Acute suicidal tendency;
4. Allergy to adhesive tape and fear of intradermal acupuncture;
5. Pregnancy and lactation;
6. Mental retardation and difficult to cooperate with doctors.
7. Participating in other clinical trials.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Changes in the Hamilton Depression Scale-17 (HAMD-17) Scores | Baseline, 3 weeks after treatment, 6 weeks after treatment, at 4-week follow-up.
  The HAMD scale is the most commonly used in the clinical assessment of depression, including 17 items. The higher the score, the more severe the depression. 0-7 means no depressive symptoms, 8-17 means mild depression, 18-24 was divided into moderate depression, and 25-52 was divided into severe depression.

SECONDARY OUTCOMES:
Changes in the Self-Rating Depression Scale (SDS) Scores | Baseline, 3 weeks after treatment, 6 weeks after treatment, at 4-week follow-up
  The standard score is the total of all scores multiplied by 1.25 to the nearest whole number on this scale, which has 20 questions. A standard score below 50 is normal; 50-60 is mild depression; 61-70 is moderate depression; 70 or more is severe depression.
Changes in the Pittsburgh Sleep Quality Index (PSQI) Scores | Baseline, 3 weeks after treatment, 6 weeks after treatment, at 4-week follow-up
  The PSQI is used to assess the sleep quality of the participant in the last 1 month and consisted of 19 self-rated and 5 other rated items. The higher the score, the worse the sleep quality. Sleep quality is divided into 4 levels according to the total score.
Changes in the Treatment Emergent Symptom Scale (TESS) Scores | Baseline, 6 weeks after treatment
  The TESS is often used to assess the side effects of drugs. It contains 35 symptom items and 2 total assessment items, including behavioural toxicity, laboratory tests, autonomic nervous system, nervous and cardiovascular system, etc. Each of these symptoms is graded into 5 levels of severity (0-4), with the higher the score the more severe the side effects.
Adverse Events | Up to 10 weeks
  Adverse events such as bleeding, haematoma, or unbearable pain caused by the needle, as well as drug-induced nausea, vomiting or dizziness, will all be recorded.

OTHER OUTCOMES:
Magnetic resonance imaging (MRI) data acquisition | Baseline, 6 weeks after treatment
  Brain MRI will be taken by the 3.0 T magnetic resonance scanner to analyse the functional connectivity of the patient's brain regions, particularly the hypothalamus, before and after the intervention.
Magnetic resonance spectroscopy (MRS ) data acquisition | Baseline, 6 weeks after treatment
  MRS will be taken by the 3.0 T magnetic resonance scanner to detect the neurometabolic change in patients' brain regions, particularly the hypothalamus, before and after the intervention.
Blood samples biobank establishment | Baseline, 6 weeks after treatment
  Blood samples will be collected to test the function of the hypothalamic-pituitary-adrenal axis, including the level of adrenocorticotropic hormone (ACTH) and cortisol (Cor).

CONTACTS AND LOCATIONS:
Overall Officials: Xiaomei Shao, Ph.D, Principal Investigator — The Third Affiliated hospital of Zhejiang Chinese Medical University
Locations (1):
- the Third affiliated hospital of Zhejiang Chinese Medical university, Hangzhou, Zhejiang, China